CLINICAL TRIAL: NCT03491176
Title: Quantification of Tumor Imaging Kinetics and Blood Biomarkers in Head and Neck Cancer Patients
Brief Title: Magnetic Resonance (MR) Imaging & Blood Biomarkers for Head and Neck Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA16-1041; NCI-2018-02631 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA16-1041 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-03-23; First posted 2018-04-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Squamous Cell Carcinoma of the Head and Neck; Healthy Subject; Head and Neck Cancer
Keywords: Head and Neck Cancer; Magnetic resonance imaging; MRI; Biomarker testing; Blood draws; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic (MRI, blood sample collection): Patients undergo MRI scans and collection of blood samples for biomarker testing pre-radiation therapy, weekly during radiation therapy, and at 2-3 months post-radiation therapy.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Procedure: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The goal of this research study is to find out if using additional MRIs and biomarker testing can help researchers learn to predict how the tumor may change during radiation therapy.

Biomarkers are found in the blood/tissue and may be related to participant's reaction to treatment. Biomarker testing in the study may include genetic biomarkers.

This is an investigational study. MRIs on this study are performed using FDA-approved and commercially available methods. Having added scans and blood tests is investigational.

Up to 100 participants will be enrolled in this study (up to 80 patients and up to 20 healthy volunteers in another part of the study). All will take part at MD Anderson.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the prognostic value of pretreatment volumetric tumor growth velocity (TGV), weekly tumor kinetics (TK), and blood biomarkers of mucosal head and neck cancers during radiation therapy (RT), using magnetic resonance imaging (MRI).

SECONDARY OBJECTIVES:

I. To assess functional imaging kinetics as a marker of tumor locoregional control.

II. To correlate blood biomarkers with tumor kinetics during treatment. III. To generate preliminary data for future trials.

OUTLINE:

Patients undergo MRI scans and collection of blood samples for biomarker testing pre-radiation therapy, weekly during radiation therapy, and at 2-3 months post-radiation therapy.

After completion of study, patients are followed up weekly.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven diagnosis of squamous cell carcinoma (SCC) of head and neck mucosa. Clinical evidence should be documented, and may consist of imaging, endoscopic evaluation, palpation, and should be sufficient to estimate the size of the primary for purposes of T staging
* No distant metastases, based on routine staging workup
* Consent for blood collection for biomarker analysis
* No head and neck surgery of the primary tumor or lymph nodes except for incisional or excisional biopsies
* Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2
* Dispositioned to curative intent radiotherapy
* For females of child-bearing age, a negative pregnancy test

Exclusion Criteria:

* Previous radiation treatment for head and neck mucosal primary cancers within the past 5 years (i.e. oropharynx, nasopharynx, hypopharynx, larynx, and oral cavity)
* Pregnant or breast-feeding females
* Contraindications to magnetic resonance (MR) imaging (e.g. implanted metallic prostheses, defibrillators, or stimulators)
* History of claustrophobia
* Contraindications to gadolinium contrast (e.g. kidney dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Tumor growth velocity (TGV) | Baseline and up to 2-3 months after completion of radiation therapy
  TGV is the calculated daily increase in tumor size from diagnosis to immediately before first radiotherapy (RT) treatment as measured via magnetic resonance imaging (MRI). Will use graphs and descriptive statistics to evaluate the relationship between TGV, tumor kinetics (TK), and circulating tumor cells (CTCs) with response.
Change in TK | Baseline up to 2-3 months after radiation therapy
  Tumor kinetics is the weekly decrease or increase in tumor volume after initiation of radiotherapy, evaluated using MRI. Will also use generalized linear mixed models (GLMMs) to evaluate TK over time and to assess whether a difference exists between patients with complete response (CR) and those without CR. Will use graphs and descriptive statistics to evaluate the relationship between TGV, TK, and CTCs with response.
Change in Blood Biomarkers of Mucosal Head and Neck Cancers During Radiation Therapy (RT) | Baseline and up to 2-3 months after completion radiation treatment.
  Will use GLMMs to evaluate CTCs over time and to assess whether a difference exists between patients with CR and those without CR. Will use graphs and descriptive statistics to evaluate the relationship between TGV, TK, and CTCs with response.

SECONDARY OUTCOMES:
Locoregional control | From date of first treatment to date of death, disease progression or recurrence, whichever occurs first, assessed up to 2 years
  Locoregional control is defined as 2-year disease-free survival (DFS). Proportional hazards models will be created to examine the trajectory and intercept of TK and CTCs during radiation therapy with DFS. Time-varying covariates longitudinal modeling will be used to assess the relationship between TK and CTCs.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton D Fuller, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ng SP, Bahig H, Wang J, Cardenas CE, Lucci A, Hall CS, Meas S, Sarli VN, Yuan Y, Urbauer DL, Ding Y, Ikner S, Dinh V, Elgohari BA, Johnson JM, Skinner HD, Gunn GB, Garden AS, Phan J, Rosenthal DI, Morrison WH, Frank SJ, Hutcheson KA, Mohamed ASR, Lai SY, Ferrarotto R, MacManus MP, Fuller CD. Predicting treatment Response based on Dual assessment of magnetic resonance Imaging kinetics and Circulating Tumor cells in patients with Head and Neck cancer (PREDICT-HN): matching 'liquid biopsy' and quantitative tumor modeling. BMC Cancer. 2018 Sep 19;18(1):903. doi: 10.1186/s12885-018-4808-5. PMID 30231854
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org